CLINICAL TRIAL: NCT05906303
Title: Caffeine in the Second Stage: A Randomized Control Trial in Low-risk Nulliparous Mothers at Term
Brief Title: Caffeine in the Second Stage of Labor in Low-risk Nulliparous Mothers at Term
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Reading Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-113
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Second Stage of Labor
MeSH Terms: interventions — caffeine, sodium benzoate drug combination; Saline Solution

STUDY DESIGN:
Intervention Model Description: Single Blind, Randomized control trial
Who Masked: Participant
Masking Description: Patient will receive either a mixture of caffeine and sodium benzoate dissolved in 500 cc normal saline or normal saline alone. A randomization schedule held by the OB team to determine which arm the patient falls into. The product will be prepared by pharmacy and sent to the labor floor. The infusion will be started once the patient is determined to be 10 cm in cervical dilation without notice to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Caffeine and sodium benzoate (Experimental): Patients will received 250 mg IV caffeine and sodium benzoate (125 mg each) dissolved in 500 cc normal saline which will be administered over the course of two hours upon determination the patient is 10 cm in cervical dilation.
  Interventions: Drug: Caffeine and Sodium Benzoate Injection
- Placebo (Placebo Comparator): Patients will received 500 cc normal saline which will be administered over the course of two hours upon determination the patient is 10 cm in cervical dilation.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Caffeine and Sodium Benzoate Injection — Provide caffeine to shorten second stage of labor and augment pushing efforts
  Arms: Caffeine and sodium benzoate
Drug: Normal Saline — Provide normal saline to serve as a placebo
  Arms: Placebo

SUMMARY:
Single blind, randomized control trial to determine benefit of caffeine and sodium benzoate on the second stage of labor

DETAILED DESCRIPTION:
Patients will present to the Women's Health Center as part of their prenatal visits or to Labor and Delivery for induction of labor or in spontaneous labor. Starting at 36 weeks gestation in the clinic or upon arrival to the labor floor, the inclusion criteria specified above will be applied by the OB Resident. Upon meeting criteria, the OB Resident will speak to the patient and gather any information typically needed for their visit/admission. Upon conclusion of the visit/admission, the OB Resident will discuss the consent form with the patient and inquire about interest to participate in the study. If interested in participation, the consent form will be signed by the patient, the resident, and a witness. At that time the patient will be designated a number for tracking purposes and a caffeine food frequency questionnaire will be completed. Patients who are involved in the study will have their problem list updated for tracking and will be designated on the labor board at time of arrival to maintain continuity of care within and across shifts. At time of arrival to the labor floor the OB resident with confirm desire to proceed with the study and record caffeine intake on the day of admission. Based on the previously assigned number, the patient will be placed into the treatment or placebo arm based upon a randomization schedule held by the OB resident team. At the time of labor, patient management will take place by the OB team with no impact by study involvement. At the time the patient is noted to be 10 cm dilated administration of either 500 cc normal saline (NS) or 250 mg of caffeine sodium benzoate (125 mg caffeine, 125 mg sodium benzoate) in 500 cc NS over 2 hours at a rate of 250 ml/hr will be performed. The time the intervention is given will be annotated on the labor board. The solutions will be kept in the hospital pharmacy and will be sent to the labor floor upon placement of the order in epic by the OB resident. The length of the second stage as well as the time and method of delivery, indication, blood loss and fetal APGARs will be documented in EPIC as part of the normal flow of documentation. All data will be extrapolated from EPIC, de-identified and stored in REDCap for organization and application of data analysis.

The intent of this project is to utilize a well-studied substance with the potential to improve cognitive and physiologic performance in a novel setting for a population that has a baseline risk for morbidity. The length of the overall labor process often results in a state of exhaustion for mothers prior to being required to spend potentially 2-4 hours actively pushing. The provision of caffeine may improve energy, mood and physiologic performance and reduce the incidence of operative deliveries, shorten the second stage of labor and reduce maternal blood loss. If the results of this study are demonstrated to be significant, the administration of caffeine is a low-risk intervention that may be considered for implementation across populations and potentially reduce maternal morbidity worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous pregnant mothers at term (37 weeks gestation and above), 18-45 years of age, intravenous access. Patients receiving prenatal care at Tower Health Obstetrical practices.

Exclusion Criteria:

* Hypertensive disorders (chronic hypertension, gestation hypertension, pre-eclampsia, HELLP syndrome; hypertension defined as a systolic blood pressure of 140 mmHg or diastolic blood pressure of 90 mmHg collected on two occasions four hours apart. Upon a new diagnosis of gestational hypertension, the patients would then be excluded. Chronic hypertensive patients are excluded by default.), significant cardiac history (history of myocardial infarction, stroke, arrhythmias, cardiomyopathy), positive drug screen on admission for cocaine or amphetamines (to be performed per hospital policy and provider discretion), fetal malpresentation, hepatic impairment to include a known history of fatty liver disease, cirrhosis or previously documented abnormal liver function testing (AST >39, ALT >52) or lack of prenatal care.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant patients
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Shortened second stage of labor | one year
  Decrease in the length of the second stage of labor compared to the placebo group
Reduction in maternal blood loss | one year
  Decrease in quantitative blood loss in the intervention group compared to placebo

SECONDARY OUTCOMES:
Incidence of operative delivery | one year
  Reduction in the incidence of operative delivery for maternal exhaustion in the intervention group
Fetal APGAR score | one year
  Evaluate improvements in fetal APGARs and incidence of apnea of prematurity

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jiang, MD, Principal Investigator — Reading Hospital Tower Health
Locations (1):
- Reading Hospital Labor & Delivery, West Reading, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No individual data to be shared

REFERENCES:
- [Background] Headaches in Pregnancy and Postpartum: ACOG Clinical Practice Guideline No. 3. Obstet Gynecol. 2022 May 1;139(5):944-972. doi: 10.1097/AOG.0000000000004766. PMID 35576364
- [Background] ACOG CommitteeOpinion No. 462: Moderate caffeine consumption during pregnancy. Obstet Gynecol. 2010 Aug;116(2 Pt 1):467-468. doi: 10.1097/AOG.0b013e3181eeb2a1. PMID 20664420
- [Background] Wikoff D, Welsh BT, Henderson R, Brorby GP, Britt J, Myers E, Goldberger J, Lieberman HR, O'Brien C, Peck J, Tenenbein M, Weaver C, Harvey S, Urban J, Doepker C. Systematic review of the potential adverse effects of caffeine consumption in healthy adults, pregnant women, adolescents, and children. Food Chem Toxicol. 2017 Nov;109(Pt 1):585-648. doi: 10.1016/j.fct.2017.04.002. Epub 2017 Apr 21. PMID 28438661
- [Background] Steinbrook RA, Garfield F, Batista SH, Urman RD. Caffeine for the prevention of postoperative nausea and vomiting. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):526-9. doi: 10.4103/0970-9185.119170. PMID 24249992
- [Background] Martin JA, Hamilton BE, Osterman MJK, Driscoll AK, Drake P. Births: Final Data for 2017. Natl Vital Stat Rep. 2018 Nov;67(8):1-50. PMID 30707672
- [Background] Yucel A, Ozyalcin S, Talu GK, Yucel EC, Erdine S. Intravenous administration of caffeine sodium benzoate for postdural puncture headache. Reg Anesth Pain Med. 1999 Jan-Feb;24(1):51-4. PMID 9952095
- [Background] Operative Vaginal Birth: ACOG Practice Bulletin, Number 219. Obstet Gynecol. 2020 Apr;135(4):e149-e159. doi: 10.1097/AOG.0000000000003764. PMID 32217976
- [Background] Zhang J, Landy HJ, Ware Branch D, Burkman R, Haberman S, Gregory KD, Hatjis CG, Ramirez MM, Bailit JL, Gonzalez-Quintero VH, Hibbard JU, Hoffman MK, Kominiarek M, Learman LA, Van Veldhuisen P, Troendle J, Reddy UM; Consortium on Safe Labor. Contemporary patterns of spontaneous labor with normal neonatal outcomes. Obstet Gynecol. 2010 Dec;116(6):1281-1287. doi: 10.1097/AOG.0b013e3181fdef6e. PMID 21099592
- [Background] Sheiner E, Sarid L, Levy A, Seidman DS, Hallak M. Obstetric risk factors and outcome of pregnancies complicated with early postpartum hemorrhage: a population-based study. J Matern Fetal Neonatal Med. 2005 Sep;18(3):149-54. doi: 10.1080/14767050500170088. PMID 16272036
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Southward K, Rutherfurd-Markwick KJ, Ali A. The Effect of Acute Caffeine Ingestion on Endurance Performance: A Systematic Review and Meta-Analysis. Sports Med. 2018 Aug;48(8):1913-1928. doi: 10.1007/s40279-018-0939-8. PMID 29876876
- [Background] Guest NS, VanDusseldorp TA, Nelson MT, Grgic J, Schoenfeld BJ, Jenkins NDM, Arent SM, Antonio J, Stout JR, Trexler ET, Smith-Ryan AE, Goldstein ER, Kalman DS, Campbell BI. International society of sports nutrition position stand: caffeine and exercise performance. J Int Soc Sports Nutr. 2021 Jan 2;18(1):1. doi: 10.1186/s12970-020-00383-4. PMID 33388079
- [Background] Song YJ, Kristal AR, Wicklund KG, Cushing-Haugen KL, Rossing MA. Coffee, tea, colas, and risk of epithelial ovarian cancer. Cancer Epidemiol Biomarkers Prev. 2008 Mar;17(3):712-6. doi: 10.1158/1055-9965.EPI-07-2511. PMID 18349292
- [Background] Rosenbloom JI, Rottenstreich A, Yagel S, Sompolinksy Y, Levin G. The length of the second stage of labor in nulliparous, multiparous, grand-multiparous, and grand-grand multiparous women in a large modern cohort. Eur J Obstet Gynecol Reprod Biol. 2020 Oct;253:273-277. doi: 10.1016/j.ejogrb.2020.08.029. Epub 2020 Aug 23. PMID 32898773